CLINICAL TRIAL: NCT04764474
Title: A Phase 1, Open-Label, Multicenter Study of HMPL-306 in Advanced Hematological Malignancies With Isocitrate Dehydrogenase (IDH) Mutations
Brief Title: A Study of HMPL-306 in Advanced Hematological Malignancies With mIDH
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated based on strategic evaluation of the clinical development of HMPL-306 with no safety concerns
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-306-GLOB1
Record Dates: First submitted 2021-01-19; First posted 2021-02-21 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Isocitrate Dehydrogenase Gene Mutation
Keywords: Acute Myeloid Leukemia; IDH Mutation
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): All patients will be administered HMPL-306 orally QD
  Interventions: Drug: HMPL-306

INTERVENTIONS:
Drug: HMPL-306 — Administered orally QD in a 28-day continuous dosing treatment cycle

SUMMARY:
An open label single-arm clinical trial to evaluate the safety, tolerability, PK, PD, and preliminary efficacy of HMPL-306 in subjects with advanced relapsed, refractory, or resistant hematological malignancies that harbor IDH mutations.

DETAILED DESCRIPTION:
HMPL-306 is a dual IDH1/2 inhibitor

This is a phase 1, open-label, multicenter, single-arm study to evaluate safety, tolerability, PK, PD, and preliminary efficacy of HMPL-306 administered orally in treatment of subjects with advanced relapsed, refractory, or resistant hematological malignancies that harbor IDH mutations (or co-mutations).

The study consists of 2 parts: a dose-escalation part (Part 1) and a dose-expansion part (Part 2). The dose-escalation part will determine the MTD/R2PD. The dose-expansion part will administer the MTD/RP2D to subjects with mIDH-positive AML

ELIGIBILITY:
Key Inclusion Criteria:

Subjects may be enrolled in this study only if they satisfy all the following criteria (NOTE: This is not an exhaustive list):

* Subjects aged ≥18 years.
* ECOG performance status ≤ 2
* Subjects with advanced relapsed, refractory, or resistant hematological malignancies, as defined below:

Part 1:

* Subjects with documented IDH mutation per local or institutional next generation sequence (NGS).
* Subjects must be refractory to or intolerant of established therapies.
* Subjects who have received prior IDH inhibitor treatment may be enrolled in the escalation phase.

Part 2:

* Subjects with documented IDH mutation of any of these subsets: IDH1 (R132C), IDH1 (R132H), IDH (R140Q), and IDH2 (R172K), including co-mutations and any combination thereof per local and institutional NGS.
* Patients must have received at least 1 prior line of therapy with an IDH inhibitor. An established standard of care with proven benefit for which the patient is eligible, must not be available at the time of enrollment.
* Patients with AML must not have standard therapeutic options available (including IDH inhibitors where approved) and have the following:

  * i. Relapsed AML unsuitable for intensive chemotherapy or venetoclax-based regimen or target agents;
  * ii. Primary refractory AML unsuitable for intensive chemotherapy or venetoclax-based regimen or target agents.
  * iii. Relapsed/refractory AML that has progressed on prior IDH treatment

Key Exclusion Criteria:

Subjects are not eligible for enrollment into this study if they meet any of the following criteria (NOTE: This is not an exhaustive list):

* Subjects who received an investigational agent <14 days prior to their first day of study drug administration.
* Subjects who are pregnant or breastfeeding.
* Subjects with an active severe infection, some treated infections and with an expected or with an unexplained fever >38.3°C during screening visits or on their first day of study drug administration.
* Subjects with some current or prior heart conditions.
* Subjects taking medications that are known to prolong the QT interval may not be eligible.
* Subjects with immediately life-threatening, severe complications of leukemia such as uncontrolled bleeding, pneumonia with hypoxia or shock, and/or disseminated intravascular coagulation.
* Some subjects with some current or prior gastrointestinal or liver diseases.
* Subjects with inadequate organ function as defined by the protocol.
* Subjects with a medical condition, physical examination finding, or clinical laboratory finding that, in the Investigators opinion, contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the subject at high risk from treatment complications.
* Subjects with a known hypersensitivity to HMPL-306 or to any of its excipients.
* Subjects with presence of second primary malignant tumors within the last 2 years, with the exception of the following, if medically controlled: basal cell carcinoma of the skin, squamous cell carcinoma of the skin, carcinoma in situ of the cervix, and carcinoma in situ of the breast.
* Part 2 Only: The time since the last dose of prior IDH inhibitor treatment is within 30 days prior to the first day of study drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bo Zhang, Study Director — Hutchison Medipharma Limited
Locations (15):
- United States (7):
  - University of California Irvine Medical Center (UCIMC) - Chao Family Comprehensive Cancer Center, Orange, California
  - Winship Cancer Institute - Emory University, Atlanta, Georgia
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Froedtert-Medical College of WI, Milwaukee, Wisconsin
- Spain (8):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario La Fe, Valencia, Valencia
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Institut Catala d'Oncologia de l'Hospitalet de Llobregat - Hospital Duran i Reynals, Barcelona
  - START Madrid - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 1, 2-part, open-label study was conducted in patients with advanced relapsed/refractory or resistant hematological malignancies that harbor isocitrate dehydrogenase mutations. The study consisted of dose escalation part (Part 1) and dose expansion part (Part 2). A total of 46 patients were enrolled in this study.
Pre-assignment Details: As only 1 patient was enrolled in dose expansion part, all data of patient were pooled in dose escalation part at Dose Level 8 cohort (Cohort 8) for the data analysis. Thus, no separate participant flow period was created for dose expansion part. Study was terminated based on strategic evaluation of clinical development of HMPL-306 with no safety concerns. Dose levels increase from 1 to 8, with Dose Level 1 being the lowest dose and Dose Level 8 the highest dose.
Groups:
- Cohort 1: HMPL-306 Dose Level 1: Patients received HMPL-306 Dose Level 1 tablet orally once on Day 1 of the pharmacokinetic (PK) week (7 days prior to Cycle 1 Day 1) (applicable for dose escalation part) and then once daily (QD) from Cycle 1 Day 1 until disease progression (PD), death, intolerable toxicity, withdrawal of consent, lost to follow-up, meeting conditions for treatment discontinuation specified in protocol, or end of study, whichever came first. Each cycle duration was 28 days.
- Cohort 2: HMPL-306 Dose Level 2: Patients received HMPL-306 Dose Level 2 tablet orally once on Day 1 of the PK week (7 days prior to Cycle 1 Day 1) (applicable for dose escalation part) and then QD from Cycle 1 Day 1 until PD, death, intolerable toxicity, withdrawal of consent, lost to follow-up, meeting conditions for treatment discontinuation specified in protocol, or end of study, whichever came first. Each cycle duration was 28 days.
- Cohort 3: HMPL-306 Dose Level 3: Patients received HMPL-306 Dose Level 3 tablet orally once on Day 1 of the PK week (7 days prior to Cycle 1 Day 1) (applicable for dose escalation part) and then QD from Cycle 1 Day 1 until PD, death, intolerable toxicity, withdrawal of consent, lost to follow-up, meeting conditions for treatment discontinuation specified in protocol, or end of study, whichever came first. Each cycle duration was 28 days.
- Cohort 4: HMPL-306 Dose Level 4: Patients received HMPL-306 Dose Level 4 tablet orally once on Day 1 of the PK week (7 days prior to Cycle 1 Day 1) (applicable for dose escalation part) and then QD from Cycle 1 Day 1 until PD, death, intolerable toxicity, withdrawal of consent, lost to follow-up, meeting conditions for treatment discontinuation specified in protocol, or end of study, whichever came first. Each cycle duration was 28 days.
- Cohort 5: HMPL-306 Dose Level 5: Patients received HMPL-306 Dose Level 5 tablet orally once on Day 1 of the PK week (7 days prior to Cycle 1 Day 1) (applicable for dose escalation part) and then QD from Cycle 1 Day 1 until PD, death, intolerable toxicity, withdrawal of consent, lost to follow-up, meeting conditions for treatment discontinuation specified in protocol, or end of study, whichever came first. Each cycle duration was 28 days.
- Cohort 6: HMPL-306 Dose Level 6: Patients received HMPL-306 Dose Level 6 tablet orally once on Day 1 of the PK week (7 days prior to Cycle 1 Day 1) (applicable for dose escalation part) and then QD from Cycle 1 Day 1 until PD, death, intolerable toxicity, withdrawal of consent, lost to follow-up, meeting conditions for treatment discontinuation specified in protocol, or end of study, whichever came first. Each cycle duration was 28 days.
- Cohort 7: HMPL-306 Dose Level 7: Patients received HMPL-306 Dose Level 7 tablet orally once on Day 1 of the PK week (7 days prior to Cycle 1 Day 1) (applicable for dose escalation part) and then QD from Cycle 1 Day 1 until PD, death, intolerable toxicity, withdrawal of consent, lost to follow-up, meeting conditions for treatment discontinuation specified in protocol, or end of study, whichever came first. Each cycle duration was 28 days.
- Cohort 8: HMPL-306 Dose Level 8: Patients received HMPL-306 Dose Level 8 tablet orally once on Day 1 of the PK week (7 days prior to Cycle 1 Day 1) (applicable for dose escalation part) and then QD from Cycle 1 Day 1 until PD, death, intolerable toxicity, withdrawal of consent, lost to follow-up, meeting conditions for treatment discontinuation specified in protocol, or end of study, whichever came first. Each cycle duration was 28 days.
Period: Overall Study
Arm/Group | Cohort 1: HMPL-306 Dose Level 1 | Cohort 2: HMPL-306 Dose Level 2 | Cohort 3: HMPL-306 Dose Level 3 | Cohort 4: HMPL-306 Dose Level 4 | Cohort 5: HMPL-306 Dose Level 5 | Cohort 6: HMPL-306 Dose Level 6 | Cohort 7: HMPL-306 Dose Level 7 | Cohort 8: HMPL-306 Dose Level 8
Started | 3 | 3 | 11 | 7 | 6 | 4 | 4 | 8 (1 patient was enrolled in dose expansion part at Dose Level 8 and all data of this patient were pooled in the dose escalation part at Dose Level 8 cohort (Cohort 8) for data analysis.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 11 | 7 | 6 | 4 | 4 | 8
Not completed — Death | 1 | 3 | 7 | 5 | 5 | 3 | 2 | 4
Not completed — Sponsor terminated study | 0 | 0 | 4 | 1 | 1 | 0 | 1 | 3
Not completed — Withdrawal of consent | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all enrolled patients who received at least 1 dose of study drug.
Groups:
- Cohort 1: HMPL-306 Dose Level 1: Patients received HMPL-306 Dose Level 1 tablet orally once on Day 1 of the PK week (7 days prior to Cycle 1 Day 1) (applicable for dose escalation part) and then QD from Cycle 1 Day 1 until PD, death, intolerable toxicity, withdrawal of consent, lost to follow-up, meeting conditions for treatment discontinuation specified in protocol, or end of study, whichever came first. Each cycle duration was 28 days.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: HMPL-306 Dose Level 1 | Cohort 2: HMPL-306 Dose Level 2 | Cohort 3: HMPL-306 Dose Level 3 | Cohort 4: HMPL-306 Dose Level 4 | Cohort 5: HMPL-306 Dose Level 5 | Cohort 6: HMPL-306 Dose Level 6 | Cohort 7: HMPL-306 Dose Level 7 | Cohort 8: HMPL-306 Dose Level 8 | Total
Number analyzed (Participants) | 3 | 3 | 11 | 7 | 6 | 4 | 4 | 8 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (5.69) | 65.0 (10.15) | 72.3 (6.92) | 68.7 (5.68) | 69.2 (12.04) | 66.5 (17.71) | 67.3 (10.90) | 70.4 (13.46) | 69.2 (9.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 6 | 2 | 3 | 1 | 2 | 4 | 21
  Male | 1 | 2 | 5 | 5 | 3 | 3 | 2 | 4 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 5 | 1 | 1 | 0 | 3 | 13
  Not Hispanic or Latino | 3 | 1 | 8 | 2 | 5 | 3 | 4 | 5 | 31
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  White | 3 | 2 | 8 | 7 | 5 | 4 | 4 | 7 | 40
  Unknown or Not Reported | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation Part: Recommended Phase 2 Dose (RP2D) of HMPL-306
Description: RP2D determination took the following criteria under consideration: determination of maximum tolerated dose (MTD) achieved during the dose escalation part and assessment of safety, PK and pharmacodynamics (PD).
Time Frame: From the first dose of study drug (Day 1) up to Day 28 of Cycle 1
Population: The safety analysis set included all enrolled patients who received at least 1 dose of study drug.
Measure: Number; unit: mg
Groups:
- Dose Escalation Part: Cohorts 1 to 8: HMPL-306: All patients enrolled in the dose escalation part (Cohorts 1 to 8) were included in this arm.
Arm/Group | Dose Escalation Part: Cohorts 1 to 8: HMPL-306
Number analyzed (Participants) | 45
mg | NA — The MTD was not reached up to the explored highest dose of Dose Level 8 and the RP2D was not determined in the study.

2. Primary Outcome: Dose Escalation Part: Number of Patients With Dose-Limiting Toxicities (DLTs)
Description: DLT was defined as occurrence of any of the following treatment-emergent adverse events (TEAEs) during the DLT assessment window, unless clearly unrelated to the study drug as per investigator's discretion: nonhematologic toxicity: TEAEs of Grade >=4, Grade >=3 with the exception of those that resolved within 72 hours (h) of onset; hematologic toxicity with the exception of neutropenia or thrombocytopenia that occurred with active leukemic disease: Grade 3 or 4 neutropenia lasting more than 7 days, Grade 4 thrombocytopenia or Grade 3 thrombocytopenia with bleeding or any requirement for platelets (PLT) transfusion, Grade 3 or greater febrile neutropenia defined as absolute neutrophil count (ANC) 1000 per cubic millimeter with a single temperature of >38.3 degree Celsius (°C) or a sustained temperature of >=38°C for more than 1 h; any TEAE requiring a dose delay of >=14 days or cases of confirmed Hy's law.
Time Frame: From the first dose of study drug (Day 1) up to Day 28 of Cycle 1
Population: The DLT-evaluable analysis set included all patients provided by HUTCHMED clinical team based on the decision made with the safety review committee (SRC) after SRC meeting for each cohort during the dose escalation part. A patient was DLT-evaluable if the patient had received at least 75% of the assigned dose of study drug during the DLT assessment window or had not completed DLT assessment period due to a DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: HMPL-306 Dose Level 1 | Cohort 2: HMPL-306 Dose Level 2 | Cohort 3: HMPL-306 Dose Level 3 | Cohort 4: HMPL-306 Dose Level 4 | Cohort 5: HMPL-306 Dose Level 5 | Cohort 6: HMPL-306 Dose Level 6 | Cohort 7: HMPL-306 Dose Level 7 | Cohort 8: HMPL-306 Dose Level 8
Number analyzed (Participants) | 3 | 3 | 9 | 5 | 3 | 3 | 3 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Patients With Treatment-Emergent Adverse Events and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: AE:unfavorable and unintended sign,symptom or disease temporally associated with use of study drug or other protocol-imposed intervention, whether or not considered related to study drug. SAE:AE that resulted in death,life-threatening AE,inpatient hospitalization/prolongation of existing hospitalization,persistent/significant incapacity or substantial disruption of ability to conduct normal life functions, abnormal pregnancy outcome in child born to female patient or female partner of male patient exposed to study drug or was important medical event that jeopardized patient and required medical/surgical intervention to prevent above outcome. TEAE:AE with onset on/after start of study drug until 30 days after last dose or prior to start of subsequent anti-tumor therapy, or AE with onset before start of study drug but worsened in severity after study drug administration, or AE onset after 30 days after last dose or after start of subsequent anti-tumor therapy and treatment-related SAEs.
Time Frame: From the first dose of study drug (Day 1) up to 30 days after the last dose of study drug, approximately 25.25 months
Population: The safety analysis set included all enrolled patients who received at least 1 dose of study drug. As only 1 patient was enrolled in dose expansion part, all data of patient were pooled in dose escalation part at Dose Level 8 cohort (Cohort 8) for the data analysis. Thus, no separate arm was created for dose expansion part.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: HMPL-306 Dose Level 1 | Cohort 2: HMPL-306 Dose Level 2 | Cohort 3: HMPL-306 Dose Level 3 | Cohort 4: HMPL-306 Dose Level 4 | Cohort 5: HMPL-306 Dose Level 5 | Cohort 6: HMPL-306 Dose Level 6 | Cohort 7: HMPL-306 Dose Level 7 | Cohort 8: HMPL-306 Dose Level 8
Number analyzed (Participants) | 3 | 3 | 11 | 7 | 6 | 4 | 4 | 8
Participants
  Any TEAE | 3 | 3 | 11 | 7 | 6 | 3 | 4 | 8
  Any TESAE | 3 | 1 | 6 | 5 | 5 | 3 | 4 | 5

4. Secondary Outcome: Number of Patients With Best Overall Response (BOR)
Description: BOR was defined as the best response during the anti-tumor evaluation period, which was determined using time point responses (TPRs) from date of the first dose of study drug from Cycle 1 in continuous cycle up until the last evaluable TPR prior to or on the date of PD/relapse according to the 2017 European LeukemiaNet criteria, or death; or withdrawal of consent or lost to follow-up; or receiving subsequent anti-cancer therapy, whichever was earlier. Number of patients with BOR [complete response (CR), CR with negative minimal residual disease (CRmrd-), CR with partial hematological recovery (CRh), CR with incomplete count (CRi), morphologic leukemia-free state (MLFS), partial response (PR), stable disease (SD), and PD] are reported.
Time Frame: Tumor assessments performed every 8 weeks (+/-7 days) for the first 24 weeks and every 12 weeks (+/-14 days) thereafter until end of treatment, or end of efficacy follow-up period, approximately 45 months
Population: The efficacy analysis set included all enrolled patients who received at least 1 dose of study drug from Cycle 1 Day 1 in continuous cycle (i.e., excluding single oral dose from the PK week for the dose escalation part). As only 1 patient was enrolled in dose expansion part, all data of patient were pooled in dose escalation part at Dose Level 8 cohort (Cohort 8) for the data analysis. Thus, no separate arm was created for dose expansion part.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: HMPL-306 Dose Level 1 | Cohort 2: HMPL-306 Dose Level 2 | Cohort 3: HMPL-306 Dose Level 3 | Cohort 4: HMPL-306 Dose Level 4 | Cohort 5: HMPL-306 Dose Level 5 | Cohort 6: HMPL-306 Dose Level 6 | Cohort 7: HMPL-306 Dose Level 7 | Cohort 8: HMPL-306 Dose Level 8
Number analyzed (Participants) | 3 | 3 | 10 | 5 | 5 | 4 | 3 | 8
Participants
  CRmrd- | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  CR | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 3
  CRh | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
  CRi | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 1
  MLFS | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SD | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
  PD | 0 | 1 | 3 | 2 | 2 | 2 | 1 | 2
  Not evaluable | 2 | 2 | 1 | 1 | 0 | 1 | 0 | 1

5. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of patients with BOR being CRmrd-, CR, CRh, CRi, MLFS or PR. CR: myeloblast <5%, blast cells without Auer bodies, no blast cells in peripheral blood, no extramedullary lesion, ANC >=1.0x10^9/L, PLT >=100x10^9/L. CRmrd-: CR with negative RT-qPCR or CR with negative MFC. CRi: met all other criteria of CR but ANC <1.0x10^9/L or PLT <100x10^9/L. MLFS: myeloblast <5%, blast cells without Auer bodies, no extramedullary lesion, no hematological recovery requirements. PR: met all hematological criteria for CR, percentage of myeloblasts decreased from baseline by least 50% and reached 5% to 25%.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Cohort 1: HMPL-306 Dose Level 1 | Cohort 2: HMPL-306 Dose Level 2 | Cohort 3: HMPL-306 Dose Level 3 | Cohort 4: HMPL-306 Dose Level 4 | Cohort 5: HMPL-306 Dose Level 5 | Cohort 6: HMPL-306 Dose Level 6 | Cohort 7: HMPL-306 Dose Level 7 | Cohort 8: HMPL-306 Dose Level 8
Number analyzed (Participants) | 3 | 3 | 10 | 5 | 5 | 4 | 3 | 8
percentage of patients | 0 [NA to NA] — NA indicates that upper and lower limits of 95% confidence interval (CI) were not estimable as there were no patients with CRmrd-, CR, CRh, CRi, MLFS or PR at study termination. | 0 [NA to NA] — NA indicates that upper and lower limits of 95% CI were not estimable as there were no patients with CRmrd-, CR, CRh, CRi, MLFS or PR at study termination. | 50.0 [18.7 to 81.3] | 40.0 [5.3 to 85.3] | 60.0 [14.7 to 94.7] | 0 [NA to NA] — NA indicates that upper and lower limits of 95% CI were not estimable as there were no patients with CRmrd-, CR, CRh, CRi, MLFS or PR at study termination. | 66.7 [9.4 to 99.2] | 62.5 [24.5 to 91.5]

6. Secondary Outcome: Time to Objective Response (TTOR)
Description: TTOR was defined as the time from the date of first study drug administration from Cycle 1 in continuous cycle to the date of first objective response (CRmrd-, CR, CRh, CRi, MLFS, or PR). CR: myeloblast <5%, blast cells without Auer bodies, no blast cells in peripheral blood, no extramedullary lesion, ANC >=1.0x10^9/L, PLT >=100x10^9/L. CRmrd-: CR with negative RT-qPCR or CR with negative MFC. CRi: met all other criteria of CR but ANC <1.0x10^9/L or PLT <100x10^9/L. MLFS: myeloblast <5%, blast cells without Auer bodies, no extramedullary lesion, no hematological recovery requirements. PR: met all hematological criteria for CR, percentage of myeloblasts decreased from baseline by least 50% and reached 5% to 25%.
Time Frame: as for outcome 4
Population: Efficacy analysis set included all enrolled patients who received at least 1 dose of study drug from Cycle 1 Day 1 in continuous cycle (i.e., excluding single oral dose from PK week for dose escalation part). As only 1 patient was enrolled in dose expansion part, all data of patient were pooled in dose escalation part at Dose Level 8 cohort (Cohort 8) for the data analysis. Thus, no separate arm was created for dose expansion part. Only patients with objective response were included in analysis.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1: HMPL-306 Dose Level 1 | Cohort 2: HMPL-306 Dose Level 2 | Cohort 3: HMPL-306 Dose Level 3 | Cohort 4: HMPL-306 Dose Level 4 | Cohort 5: HMPL-306 Dose Level 5 | Cohort 6: HMPL-306 Dose Level 6 | Cohort 7: HMPL-306 Dose Level 7 | Cohort 8: HMPL-306 Dose Level 8
Number analyzed (Participants) | 0 | 0 | 5 | 2 | 3 | 0 | 2 | 5
months |  |  | 3.680 [3.09 to 5.45] | 2.316 [0.95 to 3.68] | 4.600 [1.77 to 4.90] |  | 2.891 [2.07 to 3.71] | 1.87 [1.84 to 1.87]

7. Secondary Outcome: Duration of Objective Response (DoOR)
Description: DoOR was defined as the time from the first occurrence of objective response (CRmrd-, CR, CRh, CRi, MLFS, or PR) until PD, relapse, or death due to any cause, whichever came first. CR: myeloblast <5%, blast cells without Auer bodies, no blast cells in peripheral blood, no extramedullary lesion, ANC >=1.0x10^9/L, PLT >=100x10^9/L. CRmrd-: CR with negative RT-qPCR or CR with negative MFC. CRi: met all other criteria of CR but ANC <1.0x10^9/L or PLT <100x10^9/L. MLFS: myeloblast <5%, blast cells without Auer bodies, no extramedullary lesion, no hematological recovery requirements. PR: met all hematological criteria for CR, percentage of myeloblasts decreased from baseline by least 50% and reached 5% to 25%.
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: HMPL-306 Dose Level 1 | Cohort 2: HMPL-306 Dose Level 2 | Cohort 3: HMPL-306 Dose Level 3 | Cohort 4: HMPL-306 Dose Level 4 | Cohort 5: HMPL-306 Dose Level 5 | Cohort 6: HMPL-306 Dose Level 6 | Cohort 7: HMPL-306 Dose Level 7 | Cohort 8: HMPL-306 Dose Level 8
Number analyzed (Participants) | 0 | 0 | 5 | 2 | 3 | 0 | 2 | 5
months |  |  | 5.19 [1.87 to NA] — NA indicates that upper limit of 95% CI was not estimable due to insufficient number of patients with events at study termination. | 15.28 [7.43 to NA] — NA indicates that upper limit of 95% CI was not estimable due to insufficient number of patients with events at study termination. | 0.84 [0.69 to NA] — NA indicates that upper limit of 95% CI was not estimable due to insufficient number of patients with events at study termination. |  | 1.87 [NA to NA] — NA indicates that the upper and lower limits of 95% CI were not estimable, as there were insufficient numbers of patients with 1/2 patients censored prior to any event. | 3.71 [1.87 to NA] — NA indicates that upper limit of 95% CI was not estimable due to insufficient number of patients with events at study termination.

8. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR was defined as the percentage of patients with BOR being CRmrd-, CR, CRh, CRi, MLFS, PR, or SD lasting for 3 cycles. CR: myeloblast <5%, blast cells without Auer bodies, no blast cells in peripheral blood, no extramedullary lesion, ANC >=1.0x10^9/L, PLT >=100x10^9/L. CRmrd-: CR with negative RT-qPCR or CR with negative MFC. CRi: met all other criteria of CR but ANC <1.0x10^9/L or PLT <100x10^9/L. MLFS: myeloblast <5%, blast cells without Auer bodies, no extramedullary lesion, no hematological recovery requirements. PR: met all hematological criteria for CR, percentage of myeloblasts decreased from baseline by least 50% and reached 5% to 25%. SD: Not met criteria for CR, CRi, CRmrd-, MLFS, PR, or PD.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Cohort 1: HMPL-306 Dose Level 1 | Cohort 2: HMPL-306 Dose Level 2 | Cohort 3: HMPL-306 Dose Level 3 | Cohort 4: HMPL-306 Dose Level 4 | Cohort 5: HMPL-306 Dose Level 5 | Cohort 6: HMPL-306 Dose Level 6 | Cohort 7: HMPL-306 Dose Level 7 | Cohort 8: HMPL-306 Dose Level 8
Number analyzed (Participants) | 3 | 3 | 10 | 5 | 5 | 4 | 3 | 8
percentage of patients | 33.3 [0.8 to 90.6] | 0 [NA to NA] — NA indicates that upper and lower limits of 95% CI were not estimable as there were no patients with CRmrd-, CR, CRh, CRi, MLFS, PR, or SD lasting for 3 cycles at study termination. | 60.0 [26.2 to 87.8] | 40.0 [5.3 to 85.3] | 60.0 [14.7 to 94.7] | 25.0 [0.6 to 80.6] | 66.7 [9.4 to 99.2] | 62.5 [24.5 to 91.5]

9. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the start of study drug from Cycle 1 in continuous cycle to PD, or relapse, or death due to any cause, whichever occurred first. PD was defined as increase in bone marrow blast percentage and/or absolute peripheral blood blast cells: a) myeloblasts percentage increased from baseline by >50% (if blast cells at baseline were <30%, net increased value needs to be >=15%) or myeloblasts percentage >70% continued for at least 3 months; ANC was not seen to be improved by at least 100%, reached (>0.5x10^9/L and/or PLT reached >50x10^9/L, without blood transfusion); b) the absolute peripheral blood blast cell count (WBCxblast cell ratio) increased by >50% and reached >25x10^9/L (without differentiation syndrome); or new extramedullary diseases.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: HMPL-306 Dose Level 1 | Cohort 2: HMPL-306 Dose Level 2 | Cohort 3: HMPL-306 Dose Level 3 | Cohort 4: HMPL-306 Dose Level 4 | Cohort 5: HMPL-306 Dose Level 5 | Cohort 6: HMPL-306 Dose Level 6 | Cohort 7: HMPL-306 Dose Level 7 | Cohort 8: HMPL-306 Dose Level 8
Number analyzed (Participants) | 3 | 3 | 10 | 5 | 5 | 4 | 3 | 8
months | 6.80 [NA to NA] — NA indicates that the upper and lower limits of 95% CI were not estimable, as there were insufficient numbers of patients with 2/3 patients censored prior to any event. | 3.42 [1.87 to NA] — NA indicates that upper limit of 95% CI was not estimable due to insufficient number of patients with events at study termination. | 5.08 [0.62 to NA] — NA indicates that upper limit of 95% CI was not estimable due to insufficient number of patients with events at study termination. | 7.39 [3.22 to NA] — NA indicates that upper limit of 95% CI was not estimable due to insufficient number of patients with events at study termination. | 4.57 [2.10 to NA] — NA indicates that upper limit of 95% CI was not estimable due to insufficient number of patients with events at study termination. | 3.71 [1.87 to NA] — NA indicates that upper limit of 95% CI was not estimable due to insufficient number of patients with events at study termination. | 5.55 [0.79 to NA] — NA indicates that upper limit of 95% CI was not estimable due to insufficient number of patients with events at study termination. | 4.62 [0.49 to NA] — NA indicates that upper limit of 95% CI was not estimable due to insufficient number of patients with events at study termination.

10. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the start of study drug from Cycle 1 in continuous cycle until the date of death due to any cause.
Time Frame: From the first dose of study drug (Day 1) up to date of death due to any cause, approximately 45 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: HMPL-306 Dose Level 1 | Cohort 2: HMPL-306 Dose Level 2 | Cohort 3: HMPL-306 Dose Level 3 | Cohort 4: HMPL-306 Dose Level 4 | Cohort 5: HMPL-306 Dose Level 5 | Cohort 6: HMPL-306 Dose Level 6 | Cohort 7: HMPL-306 Dose Level 7 | Cohort 8: HMPL-306 Dose Level 8
Number analyzed (Participants) | 3 | 3 | 10 | 5 | 5 | 4 | 3 | 8
months | 6.80 [NA to NA] — NA indicates that the upper and lower limits of 95% CI were not estimable, as there were insufficient numbers of patients with 2/3 patients censored prior to any event. | 4.57 [3.42 to NA] — NA indicates that upper limit of 95% CI was not estimable due to insufficient number of patients with events at study termination. | 13.01 [0.62 to NA] — NA indicates that upper limit of 95% CI was not estimable due to insufficient number of patients with events at study termination. | 15.24 [5.19 to NA] — NA indicates that upper limit of 95% CI was not estimable due to insufficient number of patients with events at study termination. | 7.66 [5.36 to NA] — NA indicates that upper limit of 95% CI was not estimable due to insufficient number of patients with events at study termination. | 9.89 [3.06 to NA] — NA indicates that upper limit of 95% CI was not estimable due to insufficient number of patients with events at study termination. | 6.01 [0.79 to NA] — NA indicates that upper limit of 95% CI was not estimable due to insufficient number of patients with events at study termination. | 13.47 [0.49 to NA] — NA indicates that upper limit of 95% CI was not estimable due to insufficient number of patients with events at study termination.

11. Secondary Outcome: Event-Free Survival (EFS)
Description: EFS was defined as the time from date of first study drug administration from Cycle 1 in continuous cycle to treatment failure, relapse from CR (including CRmrd-, CR, CRh and CRi), or death due to any cause, whichever occurred first. CR: myeloblast <5%, blast cells without Auer bodies, no blast cells in peripheral blood, no extramedullary lesion, ANC >=1.0x10^9/L, PLT >=100x10^9/L. CRmrd-: CR with negative RT-qPCR or CR with negative MFC. CRi: met all other criteria of CR but ANC <1.0x10^9/L or PLT <100x10^9/L. Treatment failure was defined as failure to achieve CR (including CRmrd-, CR, CRh, CRi) by Week 24. Patients who did not achieve CR (including CRmrd-, CR, CRh, CRi) by Week 24 were considered to have had an event at Day 1 of first study drug administration from Cycle 1 (excluding single oral dose from PK week). For remaining CR responders (including CRmrd-, CR, CRh and CRi), event time was time of either disease relapse or death due to any cause, whichever occurred first.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: HMPL-306 Dose Level 1 | Cohort 2: HMPL-306 Dose Level 2 | Cohort 3: HMPL-306 Dose Level 3 | Cohort 4: HMPL-306 Dose Level 4 | Cohort 5: HMPL-306 Dose Level 5 | Cohort 6: HMPL-306 Dose Level 6 | Cohort 7: HMPL-306 Dose Level 7 | Cohort 8: HMPL-306 Dose Level 8
Number analyzed (Participants) | 3 | 3 | 10 | 5 | 5 | 4 | 3 | 8
months | 0.03 [NA to NA] — NA indicates that the upper and lower limits of 95% CI were not estimable, as all the patients in this cohort experienced an event of treatment failure at Day 1 (0.03 months). | 0.03 [NA to NA] — NA indicates that the upper and lower limits of 95% CI were not estimable, as all the patients in this cohort experienced an event of treatment failure at Day 1 (0.03 months). | 0.03 [0.03 to 5.65] | 0.03 [0.03 to NA] — NA indicates that upper limit of 95% CI was not estimable due to insufficient number of patients with events at study termination. | 5.55 [0.03 to NA] — NA indicates that upper limit of 95% CI was not estimable due to insufficient number of patients with events at study termination. | 0.03 [NA to NA] — NA indicates that the upper and lower limits of 95% CI were not estimable, as all the patients in this cohort experienced an event of treatment failure at Day 1 (0.03 months). | 5.55 [0.03 to NA] — NA indicates that upper limit of 95% CI was not estimable due to insufficient number of patients with events at study termination. | 4.62 [0.03 to NA] — NA indicates that upper limit of 95% CI was not estimable due to insufficient number of patients with events at study termination.

12. Secondary Outcome: Number of Patients With Post-Baseline Transfusion Independence (TI)
Description: Post-baseline TI was defined as the absence of red blood cell and platelet transfusions for a pre-specified time during treatment period which was defined from the first dose of study drug administration from Cycle 1 in continuous cycle to 30 days after the last dose date or prior to the start of a subsequent anti-tumor therapy (whichever came first). Number of patients with post-baseline TI for >=4 weeks and >=8 weeks is presented.
Time Frame: From the first dose of study drug (Day 1) up to 30 days after the last dose of study drug, approximately 25.25 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: HMPL-306 Dose Level 1 | Cohort 2: HMPL-306 Dose Level 2 | Cohort 3: HMPL-306 Dose Level 3 | Cohort 4: HMPL-306 Dose Level 4 | Cohort 5: HMPL-306 Dose Level 5 | Cohort 6: HMPL-306 Dose Level 6 | Cohort 7: HMPL-306 Dose Level 7 | Cohort 8: HMPL-306 Dose Level 8
Number analyzed (Participants) | 3 | 3 | 10 | 5 | 5 | 4 | 3 | 8
Participants
  Post-baseline TI for >=4 weeks | 3 | 3 | 7 | 4 | 4 | 4 | 3 | 8
  Post-baseline TI for >=8 weeks | 0 | 0 | 6 | 2 | 4 | 1 | 2 | 6

13. Secondary Outcome: Plasma Concentrations of HMPL-306
Description: Blood samples were collected at the specified timepoints to determine plasma concentrations of HMPL-306.
Time Frame: PK Week: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 24, 48, 72, 96, 120, 144, 168 hours post-dose on Day 1 PK week; Cycle 2 Day 1: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 24 hours post-dose on Cycle 2 Day 1
Population: The PK concentration analysis set included all patients who received at least 1 dose of the study drug and had at least 1 measurable plasma concentration data point. As only 1 patient was enrolled in dose expansion part, all data of patient were pooled in dose escalation part at Dose Level 8 cohort (Cohort 8) for the data analysis. Thus, no separate arm was created for dose expansion part. Only patients with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1: HMPL-306 Dose Level 1 | Cohort 2: HMPL-306 Dose Level 2 | Cohort 3: HMPL-306 Dose Level 3 | Cohort 4: HMPL-306 Dose Level 4 | Cohort 5: HMPL-306 Dose Level 5 | Cohort 6: HMPL-306 Dose Level 6 | Cohort 7: HMPL-306 Dose Level 7 | Cohort 8: HMPL-306 Dose Level 8
Number analyzed (Participants) | 3 | 3 | 11 | 7 | 6 | 4 | 4 | 8
nanogram per milliliter (ng/mL)
  PK Week: Pre-dose on Day 1: number analyzed (Participants) | 3 | 3 | 11 | 7 | 4 | 3 | 4 | 8
  PK Week: Pre-dose on Day 1 | NA (NA) — NA indicates that mean and standard deviation (SD) were not estimable as the values were below the lower limit of quantification (LLOQ) of 1.00 ng/mL. | NA (NA) — NA indicates that mean and SD were not estimable as the values were below the LLOQ of 1.00 ng/mL. | NA (NA) — NA indicates that mean and SD were not estimable as the values were below the LLOQ of 1.00 ng/mL. | NA (NA) — NA indicates that mean and SD were not estimable as the values were below the LLOQ of 1.00 ng/mL. | NA (NA) — NA indicates that mean and SD were not estimable as the values were below the LLOQ of 1.00 ng/mL. | NA (NA) — NA indicates that mean and SD were not estimable as the values were below the LLOQ of 1.00 ng/mL. | NA (NA) — NA indicates that mean and SD were not estimable as the values were below the LLOQ of 1.00 ng/mL. | NA (NA) — NA indicates that mean and SD were not estimable as the values were below the LLOQ of 1.00 ng/mL.
  PK Week: 0.5 hour post-dose on Day 1: number analyzed (Participants) | 3 | 3 | 11 | 7 | 6 | 3 | 4 | 7
  PK Week: 0.5 hour post-dose on Day 1 | 40.6 (33.1) | 12.8 (9.02) | 155 (200) | 40.5 (66.0) | 101 (59.6) | 28.5 (41.9) | 65.0 (80.9) | 206 (266)
  PK Week: 1 hour post-dose on Day 1: number analyzed (Participants) | 3 | 3 | 11 | 7 | 5 | 4 | 4 | 7
  PK Week: 1 hour post-dose on Day 1 | 115 (67.5) | 223 (161) | 320 (256) | 249 (278) | 541 (292) | 268 (285) | 258 (171) | 826 (545)
  PK Week: 2 hours post-dose on Day 1: number analyzed (Participants) | 2 | 3 | 11 | 7 | 5 | 4 | 4 | 7
  PK Week: 2 hours post-dose on Day 1 | 151 (80.5) | 412 (260) | 417 (140) | 535 (254) | 955 (772) | 999 (112) | 777 (559) | 869 (524)
  PK Week: 3 hours post-dose on Day 1: number analyzed (Participants) | 3 | 3 | 11 | 7 | 5 | 4 | 4 | 8
  PK Week: 3 hours post-dose on Day 1 | 130 (39.5) | 275 (103) | 379 (109) | 498 (209) | 868 (853) | 970 (229) | 689 (241) | 918 (539)
  PK Week: 4 hours post-dose on Day 1: number analyzed (Participants) | 2 | 3 | 11 | 7 | 5 | 4 | 4 | 8
  PK Week: 4 hours post-dose on Day 1 | 93.9 (8.70) | 164 (64.8) | 293 (126) | 379 (114) | 596 (525) | 744 (316) | 601 (220) | 985 (703)
  PK Week: 6 hours post-dose on Day 1: number analyzed (Participants) | 3 | 3 | 11 | 7 | 6 | 3 | 3 | 8
  PK Week: 6 hours post-dose on Day 1 | 48.9 (20.6) | 131 (26.5) | 192 (76.5) | 248 (71.5) | 327 (164) | 387 (85.8) | 498 (227) | 719 (529)
  PK Week: 8 hours post-dose on Day 1: number analyzed (Participants) | 3 | 3 | 11 | 7 | 2 | 3 | 4 | 8
  PK Week: 8 hours post-dose on Day 1 | 47.3 (21.2) | 110 (32.6) | 151 (45.6) | 204 (72.5) | 249 (191) | 331 (73.7) | 375 (111) | 517 (257)
  PK Week: 24 hours post-dose on Day 1: number analyzed (Participants) | 3 | 3 | 11 | 7 | 6 | 4 | 4 | 7
  PK Week: 24 hours post-dose on Day 1 | 23.8 (2.15) | 63.5 (27.0) | 85.6 (20.6) | 113 (21.9) | 167 (76.8) | 177 (55.6) | 183 (56.6) | 301 (148)
  PK Week: 48 hours post-dose on Day 1: number analyzed (Participants) | 3 | 2 | 11 | 7 | 6 | 4 | 4 | 6
  PK Week: 48 hours post-dose on Day 1 | 17.1 (1.00) | 42.9 (23.7) | 64.3 (14.2) | 79.2 (18.4) | 119 (49.7) | 119 (22.9) | 132 (51.9) | 202 (106)
  PK Week: 72 hours post-dose on Day 1: number analyzed (Participants) | 3 | 3 | 11 | 6 | 6 | 4 | 4 | 7
  PK Week: 72 hours post-dose on Day 1 | 15.9 (3.29) | 39.9 (15.8) | 55.9 (16.1) | 66.3 (12.8) | 97.1 (48.1) | 108 (19.9) | 114 (48.4) | 167 (76.1)
  PK Week: 96 hours post-dose on Day 1: number analyzed (Participants) | 3 | 3 | 11 | 7 | 6 | 4 | 3 | 5
  PK Week: 96 hours post-dose on Day 1 | 13.4 (1.02) | 34.2 (14.9) | 52.5 (15.0) | 61.2 (11.7) | 83.8 (38.8) | 93.0 (15.3) | 88.0 (48.8) | 175 (84.6)
  PK Week: 120 hours post-dose on Day 1: number analyzed (Participants) | 2 | 3 | 10 | 7 | 5 | 4 | 4 | 6
  PK Week: 120 hours post-dose on Day 1 | 13.3 (1.56) | 32.2 (14.6) | 43.0 (13.2) | 52.9 (4.73) | 64.0 (25.9) | 79.8 (13.1) | 83.3 (38.9) | 138 (73.4)
  PK Week: 144 hours post-dose on Day 1: number analyzed (Participants) | 2 | 3 | 10 | 7 | 4 | 4 | 3 | 6
  PK Week: 144 hours post-dose on Day 1 | 11.7 (0.424) | 29.4 (12.9) | 40.5 (14.0) | 47.2 (4.18) | 56.2 (28.1) | 72.2 (3.68) | 55.8 (26.2) | 132 (71.8)
  PK Week: 168 hours post-dose on Day 1: number analyzed (Participants) | 2 | 2 | 10 | 5 | 3 | 4 | 3 | 6
  PK Week: 168 hours post-dose on Day 1 | 9.62 (0.679) | 27.6 (20.9) | 38.9 (14.8) | 46.2 (8.64) | 90.3 (24.9) | 64.6 (8.62) | 50.7 (22.7) | 125 (68.4)
  Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 1 | 2 | 5 | 4 | 4 | 3 | 2 | 6
  Cycle 2 Day 1: Pre-dose | 134 (NA) — NA indicates that SD was not estimable for only 1 patient. | 501 (244) | 765 (359) | 765 (110) | 916 (573) | 1558 (637) | 1475 (247) | 2133 (978)
  Cycle 2 Day 1: 0.5 h post-dose: number analyzed (Participants) | 1 | 2 | 6 | 4 | 2 | 3 | 2 | 5
  Cycle 2 Day 1: 0.5 h post-dose | 134 (NA) — NA indicates that SD was not estimable for only 1 patient. | 592 (404) | 921 (458) | 871 (300) | 1622 (1510) | 1632 (700) | 1585 (318) | 2616 (972)
  Cycle 2 Day 1: 1 h post-dose: number analyzed (Participants) | 1 | 2 | 7 | 4 | 2 | 3 | 2 | 5
  Cycle 2 Day 1: 1 h post-dose | 218 (NA) — NA indicates that SD was not estimable for only 1 patient. | 666 (486) | 1324 (611) | 1063 (319) | 1930 (1273) | 2167 (981) | 2250 (170) | 2776 (1066)
  Cycle 2 Day 1: 2 h post-dose: number analyzed (Participants) | 1 | 2 | 7 | 4 | 2 | 2 | 2 | 6
  Cycle 2 Day 1: 2 h post-dose | 293 (NA) — NA indicates that SD was not estimable for only 1 patient. | 755 (267) | 1191 (501) | 1208 (363) | 1910 (1075) | 2310 (919) | 2250 (594) | 3372 (948)
  Cycle 2 Day 1: 3 h post-dose: number analyzed (Participants) | 1 | 2 | 7 | 4 | 2 | 3 | 1 | 6
  Cycle 2 Day 1: 3 h post-dose | 282 (NA) — NA indicates that SD was not estimable for only 1 patient. | 738 (107) | 1084 (551) | 1227 (239) | 1730 (891) | 2213 (419) | 1630 (NA) — NA indicates that SD was not estimable for only 1 patient. | 2887 (1194)
  Cycle 2 Day 1: 4 h post-dose: number analyzed (Participants) | 2 | 2 | 7 | 4 | 2 | 3 | 2 | 6
  Cycle 2 Day 1: 4 h post-dose | 253 (89.1) | 573 (26.9) | 999 (351) | 946 (125) | 1180 (608) | 1873 (597) | 1695 (530) | 2345 (775)
  Cycle 2 Day 1: 6 h post-dose: number analyzed (Participants) | 2 | 2 | 6 | 4 | 2 | 3 | 2 | 6
  Cycle 2 Day 1: 6 h post-dose | 252 (114) | 505 (96.9) | 851 (298) | 870 (125) | 1082 (493) | 1697 (431) | 1445 (403) | 2242 (910)
  Cycle 2 Day 1: 8 h post-dose: number analyzed (Participants) | 2 | 3 | 6 | 4 | 2 | 3 | 2 | 6
  Cycle 2 Day 1: 8 h post-dose | 276 (148) | 592 (164) | 813 (397) | 829 (27.0) | 970 (523) | 1770 (502) | 1640 (636) | 2170 (972)
  Cycle 2 Day 1: 24 h post-dose: number analyzed (Participants) | 2 | 2 | 3 | 4 | 2 | 3 | 1 | 6
  Cycle 2 Day 1: 24 h post-dose | 206 (96.2) | 502 (160) | 837 (317) | 746 (96.8) | 899 (553) | 1484 (488) | 1230 (NA) — NA indicates that SD was not estimable for only 1 patient. | 2135 (1063)

14. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of HMPL-306
Description: Blood samples were collected at the specified timepoints to determine Cmax of HMPL-306.
Time Frame: as for outcome 13
Population: The PK parameters analysis set included all patients who received at least 1 dose of the study drug and had a sufficient PK profile to derive at least 1 PK parameter. As only 1 patient was enrolled in dose expansion part, all data of patient were pooled in dose escalation part at Dose Level 8 cohort (Cohort 8) for the data analysis. Thus, no separate arm was created for dose expansion part. Only patients with data collected at specified timepoints are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1: HMPL-306 Dose Level 1 | Cohort 2: HMPL-306 Dose Level 2 | Cohort 3: HMPL-306 Dose Level 3 | Cohort 4: HMPL-306 Dose Level 4 | Cohort 5: HMPL-306 Dose Level 5 | Cohort 6: HMPL-306 Dose Level 6 | Cohort 7: HMPL-306 Dose Level 7 | Cohort 8: HMPL-306 Dose Level 8
Number analyzed (Participants) | 3 | 3 | 11 | 7 | 6 | 4 | 4 | 8
ng/mL
  PK Week Day 1 | 151 (33.7) | 376 (71.8) | 476 (36.6) | 574 (44.2) | 749 (76.5) | 1095 (13.4) | 865 (53.5) | 1225 (45.0)
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 3 | 6 | 4 | 2 | 3 | 2 | 6
  Cycle 2 Day 1 | 413 (51.7) | 921 (30.2) | 1239 (61.6) | 1365 (21.6) | 1804 (70.7) | 2455 (31.1) | 2385 (16.1) | 3301 (31.5)

15. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) of HMPL-306
Description: Blood samples were collected at the specified timepoints to determine Tmax of HMPL-306.
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 1: HMPL-306 Dose Level 1 | Cohort 2: HMPL-306 Dose Level 2 | Cohort 3: HMPL-306 Dose Level 3 | Cohort 4: HMPL-306 Dose Level 4 | Cohort 5: HMPL-306 Dose Level 5 | Cohort 6: HMPL-306 Dose Level 6 | Cohort 7: HMPL-306 Dose Level 7 | Cohort 8: HMPL-306 Dose Level 8
Number analyzed (Participants) | 3 | 3 | 11 | 7 | 6 | 4 | 4 | 8
hour
  PK Week Day 1 | 1.98 [0.950 to 2.92] | 1.93 [1.83 to 3.00] | 1.98 [0.933 to 3.00] | 1.92 [1.02 to 3.00] | 2.00 [1.00 to 3.00] | 3.00 [2.23 to 4.00] | 3.06 [2.10 to 6.00] | 2.09 [1.00 to 6.05]
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 3 | 6 | 4 | 2 | 3 | 2 | 6
  Cycle 2 Day 1 | 2.38 [2.10 to 2.67] | 2.43 [1.03 to 2.98] | 1.00 [1.00 to 4.00] | 2.50 [2.00 to 3.00] | 1.50 [1.00 to 2.00] | 2.00 [1.03 to 3.00] | 1.51 [1.00 to 2.02] | 2.00 [1.92 to 2.87]

16. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From 0 to 24 Hours (AUC0-24) of HMPL-306
Description: Blood samples were collected at the specified timepoints to determine AUC0-24 of HMPL-306.
Time Frame: PK Week: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 24 hours post-dose on Day 1 PK week; Cycle 2 Day 1: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 24 hours post-dose on Cycle 2 Day 1
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort 1: HMPL-306 Dose Level 1 | Cohort 2: HMPL-306 Dose Level 2 | Cohort 3: HMPL-306 Dose Level 3 | Cohort 4: HMPL-306 Dose Level 4 | Cohort 5: HMPL-306 Dose Level 5 | Cohort 6: HMPL-306 Dose Level 6 | Cohort 7: HMPL-306 Dose Level 7 | Cohort 8: HMPL-306 Dose Level 8
Number analyzed (Participants) | 3 | 3 | 11 | 7 | 6 | 4 | 4 | 8
h*ng/mL
  PK Week Day 1 | 1143 (34.8) | 2625 (42.7) | 3780 (23.8) | 4811 (22.1) | 6436 (58.0) | 8368 (16.4) | 7846 (36.3) | 11211 (47.1)
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 3 | 6 | 4 | 2 | 3 | 2 | 6
  Cycle 2 Day 1 | 5697 (52.3) | 12904 (24.0) | 19159 (53.6) | 20313 (8.5) | 23740 (66.9) | 39882 (34.6) | 37973 (30.1) | 50156 (43.2)

17. Secondary Outcome: Maximum Inhibition Rate of Plasma 2-Hydroxyglutaric Acid (2-HG)
Description: Blood samples were collected at the specified timepoints to determine plasma concentrations of 2-HG which was a PD marker. The maximum inhibition rate for patients in different dose groups are presented.
Time Frame: From PK Week Day 2 until end of treatment, approximately 24.25 months
Population: The PD analysis set included all patients with at least 1 quantifiable level of 2-HG in plasma. As only 1 patient was enrolled in dose expansion part, all data of patient were pooled in dose escalation part at Dose Level 8 cohort (Cohort 8) for the data analysis. Thus, no separate arm was created for dose expansion part. Only patients with data collected are reported.
Measure: Mean (Standard Deviation); unit: percentage of inhibition
Arm/Group | Cohort 1: HMPL-306 Dose Level 1 | Cohort 2: HMPL-306 Dose Level 2 | Cohort 3: HMPL-306 Dose Level 3 | Cohort 4: HMPL-306 Dose Level 4 | Cohort 5: HMPL-306 Dose Level 5 | Cohort 6: HMPL-306 Dose Level 6 | Cohort 7: HMPL-306 Dose Level 7 | Cohort 8: HMPL-306 Dose Level 8
Number analyzed (Participants) | 3 | 3 | 11 | 7 | 5 | 4 | 4 | 8
percentage of inhibition | 65.85 (24.70) | 71.49 (33.07) | 61.23 (33.67) | 82.67 (14.21) | 59.51 (61.62) | 88.54 (11.11) | 94.28 (4.82) | 87.47 (13.23)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first dose of study drug (Day 1 of the PK week) up to 30 days after the last dose of study drug, or prior to the start of a subsequent anti-tumor therapy (whichever came first), approximately 25.25 months. All-cause mortality (deaths) were collected from the first dose of study drug (Day 1 of the PK week) up to end of follow-up, approximately 45 months.
Description: The safety analysis set included all enrolled patients who received at least 1 dose of study drug. As only 1 patient was enrolled in dose expansion part, all data of patient were pooled in dose escalation part at Dose Level 8 cohort (Cohort 8) for the data analysis. Thus, no separate arm was created for dose expansion part.
Arm/Group | Cohort 1: HMPL-306 Dose Level 1 | Cohort 2: HMPL-306 Dose Level 2 | Cohort 3: HMPL-306 Dose Level 3 | Cohort 4: HMPL-306 Dose Level 4 | Cohort 5: HMPL-306 Dose Level 5 | Cohort 6: HMPL-306 Dose Level 6 | Cohort 7: HMPL-306 Dose Level 7 | Cohort 8: HMPL-306 Dose Level 8
All-Cause Mortality (participants affected / at risk) | 1/3 | 3/3 | 7/11 | 5/7 | 5/6 | 3/4 | 2/4 | 4/8
Serious Adverse Events (participants affected / at risk) | 3/3 | 1/3 | 6/11 | 5/7 | 5/6 | 3/4 | 4/4 | 5/8
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 10/11 | 7/7 | 6/6 | 3/4 | 3/4 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: HMPL-306 Dose Level 1 (N=3) | Cohort 2: HMPL-306 Dose Level 2 (N=3) | Cohort 3: HMPL-306 Dose Level 3 (N=11) | Cohort 4: HMPL-306 Dose Level 4 (N=7) | Cohort 5: HMPL-306 Dose Level 5 (N=6) | Cohort 6: HMPL-306 Dose Level 6 (N=4) | Cohort 7: HMPL-306 Dose Level 7 (N=4) | Cohort 8: HMPL-306 Dose Level 8 (N=8)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 3 (6) | 1 (1) | 2 (2) | 0 (0) | 2 (4) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 2 (5) | 0 (0) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Differentiation syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulite (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: HMPL-306 Dose Level 1 (N=3) | Cohort 2: HMPL-306 Dose Level 2 (N=3) | Cohort 3: HMPL-306 Dose Level 3 (N=11) | Cohort 4: HMPL-306 Dose Level 4 (N=7) | Cohort 5: HMPL-306 Dose Level 5 (N=6) | Cohort 6: HMPL-306 Dose Level 6 (N=4) | Cohort 7: HMPL-306 Dose Level 7 (N=4) | Cohort 8: HMPL-306 Dose Level 8 (N=8)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bartholinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (10) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (2) | 3 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 2 (7) | 0 (0) | 1 (2) | 2 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 3 (7)
Increased tendency to bruise (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperleukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1) | 2 (4) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (2)
Fatigue (General disorders) | 3 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased activity (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nodule (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Puncture site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 1 (4) | 0 (0) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral blood blister (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (7) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (9) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (2) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Adjustment disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cranial nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pallor (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splinter (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Differentiation syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immunodeficiency (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated based on strategic evaluation of the clinical development of HMPL-306 with no safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-11-06): https://cdn.clinicaltrials.gov/large-docs/74/NCT04764474/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-06): https://cdn.clinicaltrials.gov/large-docs/74/NCT04764474/SAP_001.pdf